CLINICAL TRIAL: NCT00031187
Title: Phase II Study of SGN-15 (cBR96 - Doxorubicin Immunoconjugate) Combined With Taxotere in Patients With Hormone Refractory Prostate Carcinoma
Brief Title: Study of SGN-15, Antibody-Drug Conjugate, to Treat Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SG0001-015; NCT00028470 (obsolete NCT alias)
Record Dates: First submitted 2002-02-27; First posted 2002-02-28 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate; Lewis Blood-Group System; Antibodies, Monoclonal; Antigens, Neoplasm; Antineoplastic Agents
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — BR96-doxorubicin immunoconjugate; Docetaxel

INTERVENTIONS:
Drug: SGN-15 (cBR96-doxorubicin immunoconjugate)
Drug: Taxotere (docetaxel)

SUMMARY:
SGN-15 is being investigated for therapy of patients with prostate cancer in combination with the cytotoxic agent, Taxotere. The study is an open label, randomized phase II study for patients with documented hormone refractory prostate cancer who have not had any prior therapy with Taxotere or Novantrone. Both SGN-15 and Taxotere will be administered weekly over two 6 week courses separated by a 2 week rest period.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a new class of biologic agent, the monoclonal antibody (mAb) drug conjugate SGN-15 (cBR96 - Doxorubicin immunoconjugate), used in combination with the taxane agent, TAXOTERE (docetaxel) as a strategy for targeting advanced stage, hormone refractory prostate carcinoma (HRPC). This is a randomized, open label, phase II study evaluating the immunoconjugate SGN-15 in combination with the taxane TAXOTERE in comparison to TAXOTERE alone in patients with HRPC. Based on a previous phase I study of the SGN-15/TAXOTERE combination, the weekly dose of SGN-15 will be 200 mg/m2 and the weekly dose of TAXOTERE will be 35 mg/m2. The schedule of administration for both agents will be weekly, with SGN-15 administered prior to the TAXOTERE in the patients treated with the combination. A single course of therapy will be defined as 6 weekly doses followed by a 2 week rest period for a total of 8 weeks. The study will perform an interim analysis of the data after 80 patients have completed two courses. Patients should be treated for a minimum of 2 courses of therapy. Additionally, for patients who remain eligible and have experienced tolerable levels of drug toxicity, repeat dosing with subsequent cycles is possible. Patients will be removed from study if there is evidence of tumor progression or intolerable toxicity. Follow-up assessments include adverse event reporting, clinical laboratory studies, and quality of life (QOL) assessment using a validated QOL instrument.

ELIGIBILITY:
BRIEF:

Patients must have pathologically confirmed prostate cancer, which is refractory to hormone therapy. There must be evidence of advancing disease, determined by increasing bidimensional or unidimensional measurable tumor or an increasing PSA with documented metastatic disease.

Patients must have Lewis(Y) antigen expression documented by immunohistochemistry on archived or fresh tumor specimen.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2000-10; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sandler, MD, Study Director — Seagen Inc.
Locations (11):
- United States (11):
  - Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - West Los Angeles - VA Healthcare Center, Los Angeles, California
  - VA Medical Center of Palo Alto, Palo Alto, California
  - Sharp HealthCare, Sidney Kimmel Cancer Center, San Diego, California
  - Bendheim Cancer Center, Greenwich, Connecticut
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Innovative Medical Research of South Florida, Miami Shores, Florida
  - St. Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Arlington Fairfax Hematology-Oncology, P.C., Arlington, Virginia

REFERENCES:
- See also: Click here for more information about this study and the sponsor — http://www.seattlegenetics.com